CLINICAL TRIAL: NCT01040195
Title: A Prospective Double Blind Placebo Controlled Trial of Combination Disease Modifying Antirheumatic Drugs (DMARDs) vs Monotherapy (Sulfasalazine) in Patients With Inflammatory Low Backache in Early Seronegative Spondylarthropathy
Brief Title: Combination Disease-Modifying Antirheumatic Drugs (DMARDs) Versus Sulfasalazine in Inflammatory Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Vikas Agarwal, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-08:PGI/DM/IEC/45/7.2.2009
Record Dates: First submitted 2009-12-25; First posted 2009-12-29 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Seronegative Spondyloarthropathies
Keywords: ankylosing spondylitis; undifferentiated spondyloarthropathy; spondyloarthropathy; inflammatory back pain; methotrexate; sulfasalazine; hydroxychloroquine
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthropathies | interventions — Methotrexate; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination DMARD (Active Comparator): All patients included in the study, will be started on Sulfasalazine 1 gm once daily and in the absence of side effects increased to 2gm daily. All patients will also receive folic acid 5 mg thrice weekly. At the end of four weeks the patients will be reassessed with baseline hemogram, SGPT, SGOT and serum Creatinine. In the absence of any contraindication, patients will be randomized into two groups Group 1 to receive Combination Disease Modifying therapy with Sulfasalazine, Methotrexate and hydroxychloroquine (HCQ). Patient will be started on Methotrexate/placebo at 10 mg once weekly and increased every week by 2.5 mg to maximum dose of 20 mg per week in the absence of side effects. These patients will also be started on Hydroxychloroquine 200 mg per day.
  Interventions: Drug: Methotrexate, Hydroxychloroquine
- Placebo (Placebo Comparator): All patients included in the study, will be started on Sulfasalazine 1 gm once daily and in the absence of side effects increased to 2gm daily All patients will also receive folic acid 5 mg twice weekly. At the end of four weeks the patients will be reassessed with baseline hemogram, SGPT, SGOT and serum Creatinine. Group 2 patients will receive Sulfasalazine and placebo for methotrexate and hydroxychloroquine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate, Hydroxychloroquine — Methotrexate will be prepared as unmarked tablets of 2.5 mg strength each and Hydroxychloroquine as unmarked tablet of 200 mg strength. Patients will be started on Methotrexate/placebo at 10 mg once weekly and increased every week by 2.5 mg to maximum dose of 20 mg per week in the absence of side effects. These patients will also be started on Hydroxychloroquine 200 mg per day or placebo.
  Other Names: Folitrax; HCQS
  Arms: Combination DMARD
Drug: Placebo — Identical placebos (for methotrexate and hydroxychloroquine)will be prepared and prescribed in identical fashion as the methotrexate and hydroxychloroquine in the combination DMARD arm.
  Arms: Placebo

SUMMARY:
Till now no drug has been conclusively shown to affect the natural course of the inflammatory back ache in seronegative spondylarthropathies. Non-steroidal anti-inflammatory drugs (NSAIDS) have been the main stay of treatment for these diseases for long. Despite providing good pain relief, they are largely ineffective in altering the natural course of these diseases. However, very often, in spite of therapy, pain and discomfort continues in these patients with recurrent exacerbations. Other drugs have been tried in these patients.

The DMARDS (Disease Modifying Anti Rheumatic Drugs) are a group of drugs which have come into prominence following their remarkable efficacy in the management of Rheumatoid Arthritis, another chronic inflammatory autoimmune arthritis. The major drugs which come in this group are Methotrexate, Sulfasalazine, Hydroxychloroquine and Leflunomide. Of these drugs, the most well studied drug in Spondylarthropathy is Sulfasalazine. Trials have shown variable results of response of spondyloarthropathy to sulfasalazine. The other major DMARD tried is methotrexate. Though large well controlled trials are lacking, the available data on its efficacy in spondyloarthropathy has not been favorable. Leflunomide, the other major DMARD has also fared poorly in a controlled trial in ankylosing spondylitis. There is at present inadequate data regarding the efficacy of Hydroxychloroquine.

The discovery of anti TNF-α have been the major breakthrough in the management of ankylosing spondylitis (AS) and Spondyloarthropathies (SpA). These drugs, besides providing symptomatic improvement, also produce improvement in the indices of disease activity as Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and the Assessment of Spondylo-Arthritis International Society (ASAS). Besides, the enormous cost, incurred at a rate of about Rs 700,000/- per annum, put it out of reach of the majority of affected population. Add to these is the increased risk of tuberculosis and fungal infections, a major problem in India.

In this background there is severe and pressing need for alternate safe and effective drugs in the management of these diseases. It is here that the combination DMARD therapy assumes importance as a potential safe and cheaper alternative.

We aim to assess the efficacy of combination DMARD therapy in patients with early inflammatory chronic backache in patients with sero negative spondyloarthropathies.

DETAILED DESCRIPTION:
Spondyloarthropathies SpA

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled criteria for the diagnosis of Ankylosing Spondylitis (Modified New York Criteria) or undifferentiated spondyloarthropathy (UspA) (Amor criteria) and are within 8 years of disease onset with:
* Inflammatory back Pain of more than 6 months
* BASDAI ≥4 or EMS ≥45 minutes
* Have failed maximum dose of at least one NSAID for 6 weeks.

Exclusion Criteria:

* Patients with renal diseases
* patients with hepatic diseases
* Patients with severe uncorrected anemia (Hb<7gm)
* Patients previously received full dose of sulfasalazine and/or methotrexate with inadequate relief
* Pregnant or lactating females
* Malignancy or active infection
* Patient requiring and affording biologicals
* Patients who have received steroids in the past 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary end point will be number of patients attaining Assessment of spondyloarthropathy international society 20 (ASAS20) response. | 28 weeks

SECONDARY OUTCOMES:
Improvement in Bath ankylosing spondylitis disease activity index (BASDAI) | 28 weeks
Improvement in Bath ankylosing spondylitis functional index (BASFI) | 28 weeks
Improvement in Bath ankylosing spondylitis metrology index (BASMI) | 28 weeks
Improvement in Maastricht Ankylosing Spondylitis Enthesitis Index | 28 weeks
Patient pain and global assessment of disease | 28 weeks
Physician assessment of pain and global disease | 28 weeks
change in Short form 36 (SF-36) and health assessment questionnaire (HAQ) parameters | 28 weeks
improvement in erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) | 28 weeks
Reduction in non steroidal anti-inflammatory drug (NSAID) dose | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Agarwal, MD, DM, Principal Investigator — SGPGIMS
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India